CLINICAL TRIAL: NCT00935610
Title: Effect of the Cysteine-rich Whey Protein Isolate (Immunocal®) in Combination With Physical Exercise on Muscle Function, Body Composition and Inflammatory Cytokine Levels in Elderly Persons: A Randomized, Double-blind Study
Brief Title: Effect of Immunocal® With Exercise Versus Casein With Exercise on Aging Processes in Elderly Persons
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immunotec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: AGING-IMM08
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2011-06

CONDITIONS: Aging; Sarcopenia
Keywords: Elderly persons; Muscle function and strength; Body composition; Inflammatory cytokine levels; Cognitive functions; Cysteine-rich whey protein isolate; Immunocal; Resistance training; Improved muscle function; Improved quality of life; Aging processes; Quality of life
MeSH Terms: conditions — Sarcopenia | interventions — Caseins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immunocal (Active Comparator): 20g of Immunocal
  Interventions: Dietary Supplement: Immunocal; Dietary Supplement: Casein
- Casein (Placebo Comparator): 20g of Casein
  Interventions: Dietary Supplement: Immunocal; Dietary Supplement: Casein

INTERVENTIONS:
Dietary Supplement: Immunocal — 20 grams per day of Immunocal for 135 days.
Dietary Supplement: Casein — 20 grams per day for 135 days

SUMMARY:
Aging is typically associated with a decrease in skeletal muscle mass and muscle function, which contributes decisively to disability in old age and to the loss of quality of life.Resistance exercise can increase muscle strength, function and mass in older adults.

The primary aim of this study is to determine whether the combination of resistance training with a supplementation of a cysteine- rich whey protein isolate (Immunocal) compared to combination of resistance training with casein used as control (casein contains little cysteine) could have the potential to provide a synergic beneficial impact on muscle mass and function which could translate to an improved quality of life in elderly persons.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* Estimated GFR above 45ml/min
* Total bilirubin in the normal range (0.2 to 1.2 mg/dl) AST (10-35 U/L for women and 10-50 U/L for men). ALT equal to or less than 2.5 times the upper limit of normal
* BMI between 18.5-29.9 (kg)/m2
* Sedentary (< 2 hours of structured exercise)in the last 2 or 3 months
* Based on investigator judgment according to current Canadian guidelines, medical conditions such as hypertension, diabetes and hyperlipidemia have to be stable and optimally controlled before the subject starts the study.

Exclusion Criteria:

* History of angioedema or allergic reactions to any compound used in this study.
* Milk protein intolerance
* Subjects currently using N-acetylcysteine, alpha-lipoic acid supplements, or dry whey protein supplements.
* Major surgery in the year prior to testing
* Acute coronary or vascular event within the last year or progressive angina
* Stroke within the past 2 years
* Neurologist and/or orthopedic limitations
* Uncontrolled thyroid or pituitary disease
* Medication which has a major affect on cognitive function
* Signs of early dementia as assessed by Mini-Mental State Examination
* Weight loss of more than 4kg(or more than 5% body weight) over last 6 months
* Alcohol abuse
* Medication which interferes with muscle mass i.e. (corticosteroids)
* Any life threatening conditions based on Investigator judgment.
* Subjects with allergies/intolerance to soya.
* Subjects currently undergoing immunosuppressive therapy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 99 (Actual)
Dates: Start 2009-06; Primary Completion 2013-07 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The mean of percent change in muscle strength based on leg press and chest press evaluation assessed by resistance training equipment | 45, 90, 135 days

SECONDARY OUTCOMES:
The mean of percent change in muscle strength based on hand-grip dynamometer | 45, 90 and 135 days
Percent change in lean body mass evaluated by DEXA. | 40, 90 and 135 days
The change in the plasma concentrations of Tumor Necrosis Factor-alpha (TNF-alpha), interleukin-6 (IL-6), C-reactive protein (CRP), glutathione, cysteine, asparagine, leucine and albumin | 40, 90 and 135 days
The clinical assessment of subject performance status (Quality of life and cognition, Physical Performance Test (PPT)). | 40, 90 and 135 days
Insulin sensitivity evaluated by fasting plasma glucose and insulin (HOMA-IR model). | 40, 90 and 135 days
The % change in body weight. | 40, 90 and 135 days
Bone mass density | 40, 90 and 135 days
6-min walk test | 40, 90 and 135 days

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, MD. Ph.D., Principal Investigator — Institut de Recherches Cliniques de Montreal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Karelis AD, Messier V, Suppere C, Briand P, Rabasa-Lhoret R. Effect of cysteine-rich whey protein (immunocal(R)) supplementation in combination with resistance training on muscle strength and lean body mass in non-frail elderly subjects: a randomized, double-blind controlled study. J Nutr Health Aging. 2015 May;19(5):531-6. doi: 10.1007/s12603-015-0442-y. PMID 25923482